CLINICAL TRIAL: NCT01979562
Title: Knowledge of Predicting Increased Risk for an Overuse Injury in Runners Related to the Mutual Length of Femur and Tibia and the Running Style
Brief Title: Knowledge of Predicting Increased Risk for an Overuse Injury in Runners
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Northern Orthopaedic Division, Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: N-20130074
Record Dates: First submitted 2013-11-04; First posted 2013-11-08 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Overuse Injuries; Musculoskeletal Make-up in the Lower Extremities
Keywords: Overuse injury; Femur; Tibia; Running; Prevention
MeSH Terms: conditions — Cumulative Trauma Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 100 runners: Male runners between 18-60 years.

SUMMARY:
The purpose of this study is to examine the skeleton of the legs and the running style in order to predict a possible overuse injury.

DETAILED DESCRIPTION:
The running style and the training composition and the body composition are thought to have major effect on the development of overuse injuries.

To define a prevention strategy, one must have the knowledge about risk factors and causation. The training composition is very relevant clinically but the underlying factors have not been studied yet. For the present there is no scientifical evidence of a possible relation between the body composition such as the mutual length and width of femur and tibia and the development of overuse injuries.

Thus, the aim of this study is to achieve evidence-based knowledge of these factors in order to advice runners about the precautions and to avoid that people get a sedentary lifestyle.

ELIGIBILITY:
Inclusion Criteria:

* Men between 18 and 60 years
* Access to an e-mail
* Two years running experience as a minimum
* Exercises three times weekly as a minimum, on annual average or until any excessive load on the body occurs
* Experience with running machines
* A written signed statement of consent

Exclusion Criteria:

* Lack of a written signed statement of consent
* Unwillingness to keep a journal during the running exercises
* Unwillingness to register data during the follow-up period
* Injury in the lower extremities within 3 months before baseline
* The runner uses insoles or he has been through a surgical procedure in the lower extremities
* A mental disability for example dementia or challenging behaviour
* The runner plays heavy sport, cf. American College of Sports Medicine
* Unability to read or understand Danish
* Unability to cooperate

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 100 male runners from athletic associations in Northern Jutland.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Injury defined as inappropriate musculoskeletal make-up in the lower extremities | 1 year

SECONDARY OUTCOMES:
Number of kilometres spent on running each week | 1 year
Bone contact forces on the distal tibia during the stance phase of running | 1 year

OTHER OUTCOMES:
Running pace, previous injuries and pain-relieving medication | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Rene B. Korsgaard, M.Sc., Principal Investigator — Aalborg University; Sten Rasmussen, M.D., Study Director — Orthopaedic Research Unit, Aalborg University Hospital, Denmark; Michael Voigt, Prof., PhD, Study Chair — Center for Motor-Sensory Interaction, Aalborg University; Uwe Kersting, Ass.prof., Study Chair — Aalborg University; Rasmus O. Nielsen, M.Sc., Study Chair — University of Aarhus; Uffe Læssoe, Ass. prof., Study Chair — University College, Northern Jutland, Denmark
Locations (1):
- Orthopaedic Surgery Research Unit, Aalborg University Hospital, Aalborg, Northern Jutland, Denmark